CLINICAL TRIAL: NCT05023837
Title: Evaluation of the Efficacy of Immunotherapy in Uncommon Pathological Types of Lung Cancer
Brief Title: Efficacy and Safety of Immunotherapy in Non-small Cell Lung Cancer With Uncommon Histological Type
Acronym: Esporta
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Other Study IDs: Esporta
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Uncommon Pathological Types of Lung Cancer
Keywords: Uncommon pathological types of lung cancer; Immune checkpoint inhibitor
MeSH Terms: interventions — pembrolizumab; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pembrolizumab 100 MG Injection — Pembrolizumab iv 200mg q21d

SUMMARY:
This study was designed to explore the efficacy and safety of immune checkpoint inhibitor for advanced uncommon pathological types of lung cancer whether or not it is accompanied by a driver mutationin the real world. Through retrospective collection of clinical data of patients with uncommon pathological types of lung cancer.The patients who are treated with immunosuppressive agents are screened out, and they are divided into immune combination therapy or immune monotherapy, and further evaluate whether there is a difference in efficacy between the two.

DETAILED DESCRIPTION:
This is a research project involving patients in Medical Oncology Department of Affiliated Cancer Hospital of Xiangya School of Medicine Central South University. Retrospective study of 40 patients with advanced uncommon pathological types of lung cancer and observe the efficacy and safety of immune checkpoint inhibitor regimen in the real world. The patients who are treated with immunosuppressive agents are screened out, and they are divided into immune combination therapy or immune monotherapy, and further evaluate whether there is a difference in efficacy between the two. Statistical analysis is used to compare the differences between the two treatments, so that patients can better choose treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18，Advanced uncommon pathological types of lung cancer by histopathology whether or not it is accompanied by a driver mutation Treatment Plan is pembrolizumab 200mg iv q21d

Exclusion Criteria:

- Patients received antitumor treatment before Patients with contraindication of chemotherapy Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced uncommon pathological types of lung cancer by histopathology
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
PFS | may 2019- may 2021
  progression survival time

SECONDARY OUTCOMES:
OS | may 2019- may 2021
  over survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Song L, Zhou F, Xu T, Zeng L, Xia Q, Wang Z, Deng L, Li Y, Qin H, Yan H, Huang Z, Mi J, Xu Q, Yang N, Zhou C, Zhang Y. Clinical activity of pembrolizumab with or without chemotherapy in advanced pulmonary large-cell and large-cell neuroendocrine carcinomas: a multicenter retrospective cohort study. BMC Cancer. 2023 May 16;23(1):443. doi: 10.1186/s12885-023-10952-w. PMID 37189075